CLINICAL TRIAL: NCT05182567
Title: Safety, Tolerability and Immunogenicity of GLS-5310 DNA Vaccine Given as a Booster to Those Previously Vaccinated Against SARS-CoV-2
Brief Title: GLS-5310 Vaccine in Healthy Volunteers as a Booster for SARS-CoV-2 (COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GeneOne Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CoV2-008
Record Dates: First submitted 2022-01-05; First posted 2022-01-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Healthy
Keywords: Vaccine; DNA
MeSH Terms: conditions — COVID-19 | interventions — GLS-5310 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GLS-5310 ID + GeneDerm 65 kPa, 30 seconds (Experimental): GLS-5310 ID + GeneDerm administered at Visit 1
  Interventions: Drug: GLS-5310 (Group 1)
- GLS-5310 ID + GeneDerm 65 kPa, 30 seconds + GLS-5310 IN (Experimental): GLS-5310 ID + GeneDerm + GLS-5310 IN administered at Visit 1
  Interventions: Drug: GLS-5310 (Group 2)
- GLS-5310 ID + GeneDerm 65 kPa, 15 seconds (Experimental): GLS-5310 ID + GeneDerm administered at Visit 1
  Interventions: Drug: GLS-5310 (Group 3)
- GLS-5310 ID + GeneDerm 80 kPa, 30 seconds (Experimental): GLS-5310 ID + GeneDerm administered at Visit 1
  Interventions: Drug: GLS-5310 (Group 4)

INTERVENTIONS:
Drug: GLS-5310 (Group 1) — GLS-5310 DNA plasmid vaccine
  Arms: GLS-5310 ID + GeneDerm 65 kPa, 30 seconds
Drug: GLS-5310 (Group 2) — GLS-5310 DNA plasmid vaccine
  Arms: GLS-5310 ID + GeneDerm 65 kPa, 30 seconds + GLS-5310 IN
Drug: GLS-5310 (Group 3) — GLS-5310 DNA plasmid vaccine
  Arms: GLS-5310 ID + GeneDerm 65 kPa, 15 seconds
Drug: GLS-5310 (Group 4) — GLS-5310 DNA plasmid vaccine
  Arms: GLS-5310 ID + GeneDerm 80 kPa, 30 seconds

SUMMARY:
Phase I study to assess the safety, tolerability and immunogenicity of GLS-5310 DNA vaccine given as a booster to those previously vaccinated against SARS-CoV-2

DETAILED DESCRIPTION:
This Phase I, randomized, placebo-controlled study will assess the safety, tolerability, and immunogenicity of GLS-5310 DNA vaccine administered intradermally (ID) with or without concomitant intranasal (IN) administration given as a heterologous booster dose to those previously vaccinated against SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years of age
2. Able to provide informed consent
3. Able and willing to comply with study procedures and agree to refrain from obtaining a booster vaccination with a non-study vaccine through to the 1 month post-boost vaccination visit
4. For women of childbearing potential, able and willing to use an approved form of pregnancy prevention for at least 4 weeks from study drug administration
5. Completion of a prior vaccination series with either the BNT162b2, mRNA-1273, or Ad26.CoV.S vaccines, with or without subsequent booster vaccination, with most recent vaccination at least 6 months prior to study entry

Exclusion Criteria:

1. Persons with symptoms in the past 2 weeks consistent with possible acute SARS-CoV-2 infection (https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html)
2. Persons with a diagnosis of type 2 diabetes mellitus
3. Persons with a diagnosis of chronic kidney disease
4. Persons with a diagnosis of chronic obstructive pulmonary disease (COPD)
5. Persons with a diagnosis of heart conditions to include heart failure, coronary artery disease, prior heart attack, cardiomyopathy
6. Sickle cell disease
7. Current or planned pregnancy during the study
8. Currently breastfeeding
9. Administration of an investigational agent within 90 days of the GLS-5310 booster dose
10. Administration of a vaccine within 2 weeks prior to the GLS-5310 booster dose
11. Administration of immune globulin within 6 months of enrollment
12. Administration of an anti-TNFα inhibitor such as infliximab, adalimumab, etanercept, or anti-CD20 monoclonal antibody rituximab within 6 months from enrollment
13. Current daily treatment of systemic corticosteroids of 20 mg of prednisone or greater; or the equivalent dose of other systemic corticosteroids
14. Treatment within the four weeks prior to enrollment with any drug intended for the prophylaxis or treatment of COVID-19
15. Any prior treatment with an anti-SARS-CoV-2 monoclonal antibody or immune serum
16. Prior treatment with an anti-IL-6 inhibitor, anti-IL-1 inhibitor, anti-TNF monoclonal antibody, or anti-JAK inhibitor (see Appendix B exclusionary period for specific drugs)
17. History of malignancy
18. History of transplantation (any organ or bone marrow)
19. Current or planned chemotherapy treatment for hematologic or solid tumor during study period
20. History of other congenital or acquired immunodeficiency, excluding those with HIV infection who are taking highly active antiretroviral therapy and who have documentation of undetectable serum viral load and who have a CD4 count > 200 cells/μL on two measures at least 3 months apart
21. Not willing to allow storage and future use of samples for coronavirus-related research and/or vaccine development
22. Prisoner or subjects who are compulsorily detained for treatment of a psychiatric illness
23. Any illness or condition that, in the opinion of the investigator, may affect the safety of the subject or the evaluation of a study endpoint
24. History of chronic rhinosinusitis
25. History of nasal septal defect or deviated nasal septum
26. History of cleft palate
27. History of nasal polyps
28. History of other disorders that, in the opinion of the investigator, may adversely affect administration of intranasal vaccine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 48 weeks post vaccination
  Solicited/unsolicited local and systemic AEs after vaccination
Determine antibody responses after a single dose of vaccine | Through 48 weeks post vaccination
  The fold change of SARS-CoV-2 Spike binding antibodies 1-month post-booster

SECONDARY OUTCOMES:
Evaluation of positive response rate of T cell responses induced by GLS-5310 DNA vaccine | Through 48 weeks post vaccination
Evaluation of neutralizing antibody response induced by GLS-5310 relative to treatment arm | Through 48 weeks post vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Meridian Clinical Research, Rockville, Maryland
  - Meridian Clinical Research, Lincoln, Nebraska
- Clinical Research Puerto Rico, San Juan, PR, Puerto Rico